CLINICAL TRIAL: NCT02012959
Title: A Phase 3b, Multicenter, Open-label, Randomized Withdrawal Trial of the Effects of Titrated Oral SAMSCA ® (Tolvaptan) on Serum Sodium, Pharmacokinetics, and Safety in Children and Adolescent Subjects Hospitalized With Euvolemic or Hypervolemic Hyponatremia
Brief Title: Study of the Safety and Effectiveness of SAMSCA® (Tolvaptan) in Children and Adolescents With Euvolemic or Hypervolemic Hyponatremia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Issues with participant recruitment & enrollment which made the trial impossible or highly impracticable. Trial termination was not due to safety reasons.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 156-08-276; 2013-002005-59 (EudraCT Number)
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-07

CONDITIONS: Hyponatremia
Keywords: Hyponatremia; Euvolemic; Hypervolemic; Serum sodium; Dilutional hyponatremia; Electrolyte abnormality; Electrolyte imbalance; Metabolic disease
MeSH Terms: conditions — Hyponatremia; Metabolic Diseases | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolvaptan Early Withdrawal (Experimental): All participants initially received tolvaptan once daily for the first 2 days. A third day of treatment was permitted if a participant had not reached the desired sodium target improvement per the investigator's judgment.
  At the end of Day 2 (or Day 3), responders (participants who achieved an increase in serum sodium by ≥4 millimoles/liter [mmol/L]) were randomized to either the Early or Late Withdrawal Group. Non-responders could continue treatment with tolvaptan for an additional 2 days.
  Discontinued tolvaptan treatment immediately after randomization.
  All participants were observed up to 14 days post randomization.
  Interventions: Drug: Tolvaptan
- Tolvaptan Late Withdrawal (Experimental): All participants initially received tolvaptan once daily for the first 2 days. A third day of treatment was permitted if a participant had not reached the desired sodium target improvement per the investigator's judgment.
  At the end of Day 2 (or Day 3), responders (participants who achieved an increase in serum sodium by ≥4 mmol/L) were randomized to either the Early or Late Withdrawal Group in Treatment Phase B. Non-responders could continue treatment with tolvaptan for an additional 2 days.
  Continued treatment for 2 additional days.
  All participants were observed up to 14 days post randomization.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan
  Other Names: SAMSCA®

SUMMARY:
The purpose of this trial was to demonstrate that tolvaptan effectively and safely increases and maintains serum sodium concentrations in children and adolescent participants with euvolemic or hypervolemic hyponatremia.

ELIGIBILITY:
Inclusion:

* Male and female participants ≥4 weeks (or ≥44 weeks adjusted gestational age) to <18 years old
* Participants hospitalized with euvolemic or hypervolemic hyponatremia resistant to initial standard background therapy
* Persistent euvolemic or hypervolemic hyponatremia defined as being documented as <130 milliequivalent (mEq)/L and present for at least 48 hours, evidenced by at least 2 serum sodium assessments (12 hours apart)
* Ability to maintain adequate fluid intake (orally or intravenously)
* Ability to take oral medications
* Ability to comply with all requirements of the trial
* Completion of the trial-specific informed consent/assent as age appropriate
* Ability to commit to remain fully abstinent or practice double-barrier birth control as required by the trial

Exclusion:

* Evidence of hypovolemia or intravascular volume depletion
* Serum sodium <120 mEq/L
* Use of potent cytochrome P450 3A4 (CYP3A4) inhibitors in participants <12 kilogram (kg) or moderate CYP3A4 inhibitors in participants <6 kg
* Lacks free access to water (inability to respond to thirst) or without intensive care unit level fluid monitoring and management
* History or current diagnosis of nephrotic syndrome
* Transient hyponatremia likely to resolve
* Hyperkalemia
* Estimated glomerular filtration rate <30 milliliters/minute/1.73 meters squared
* Acute kidney injury
* Severe or acute neurological symptoms requiring other intervention
* Prior treatment for hyponatremia with hypertonic saline within 8 hours of qualifying serum sodium assessments; urea, lithium, demeclocycline, conivaptan, or tolvaptan within 4 days of qualifying serum sodium assessments; any other treatments for the purpose of increasing serum sodium concurrent with dosing of trial medication
* Anuria or urinary outflow obstruction, unless participant is/can be catheterized
* History of hypersensitivity and/or idiosyncratic reaction to benzazepine or benzazepine derivatives
* Psychogenic polydipsia
* Uncontrolled diabetes mellitus (defined as fasting glucose >300 milligrams/deciliter)
* Screening liver function values >3 times the upper limit of normal
* Participants who have cirrhosis and meet any of the following conditions: a major GI bleed within the past 6 months, evidence of active bleeding, platelet count <50,000/microliter, or use of concomitant medications known to increase bleeding risk
* Hyponatremia due to the result of any medication that can safely be withdrawn or that is most appropriately corrected by alternative therapies
* History of drug or medication abuse within 3 months prior to screening or current alcohol abuse
* Participants who require suspension formulation and have a Hereditary Fructose Intolerance
* Has hyponatremia that is more appropriately corrected by alternative therapies
* Is pregnant or currently breastfeeding
* Has any medical condition that could interfere with evaluation of trial objectives or participant safety
* Has participated in another investigational drug trial in the last 30 days
* Weighs <3 kg
* Unable to swallow tablets, if suspension unavailable
* Is deemed unsuitable for trial participation in the opinion of the investigator

Ages: 4 Weeks to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Development, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (7):
- United States (5):
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - New York, New York
  - Richmond, Virginia
  - Seattle, Washington
- Rome, Italy
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Phase A: During Treatment Phase A, participants received tolvaptan once daily on Days 1 and 2. If the serum sodium level did not increase at least 4 milliequivalent (mEq)/liter (L) by Day 2, treatment was extended one additional day (Day 2a). On Day 2a, participants achieving an increase in serum sodium of ≥4 mEq/L were defined as responders, and participants not achieving a ≥4 mEq/L increase in serum sodium were defined as non-responders.
- Treatment Phase B: Responder - Late Withdrawal: Participants who were responders (serum sodium increased by ≥4 mEq/L) from Phase A continued to Treatment Phase B (Randomization Phase) on Day 3 and were randomized to the Late Withdrawal group (continuing tolvaptan treatment for Days 3 and 4).
- Treatment Phase B: Responder - Early Withdrawal: Participants who were responders (serum sodium increased by ≥4 mEq/L) from Phase A continued to Treatment Phase B (Randomization Phase) on Day 3 and were randomized to the Early Withdrawal group (not receiving additional tolvaptan on Days 3 or 4). Participants randomized to Early Withdrawal were monitored for any interventions needed to maintain appropriate serum sodium levels. Where sodium levels declined by ≥4 mEq/L, or where the overall clinical condition warranted further intervention to increase serum sodium levels, participants were treated per the investigator's preferred standard of care. Any intervention, including fluid restriction, during the first 48 hours of the Early Withdrawal phase was defined as rescue therapy, and participant data was censored thereafter.
- Treatment Phase B: Non-responder - Study Drug: Participants who were non-responders during Phase A were not randomized in Phase B, but were treated per the investigator's discretion and continued tolvaptan for Days 3 and 4.
- Treatment Phase B: Non-responder - Standard of Care: Participants who were non-responders during Phase A were not randomized in Phase B, but were treated per the investigator's discretion. The participants in this arm discontinued tolvaptan and received the investigator's preferred standard of care for Days 3 and 4.
Period: Treatment Phase A
Arm/Group | Treatment Phase A | Treatment Phase B: Responder - Late Withdrawal | Treatment Phase B: Responder - Early Withdrawal | Treatment Phase B: Non-responder - Study Drug | Treatment Phase B: Non-responder - Standard of Care
Started | 9 | 0 (Zero participants noted because participants did not start Phase B yet) | 0 (Zero participants noted because participants did not start Phase B yet) | 0 (Zero participants noted because participants did not start Phase B yet) | 0 (Zero participants noted because participants did not start Phase B yet)
Received At Least 1 Dose of Study Drug (Phase A Safety Sample) | 9 | 0 | 0 | 0 | 0
Completed | 7 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0
Period: Treatment Phase B
Arm/Group | Treatment Phase A | Treatment Phase B: Responder - Late Withdrawal | Treatment Phase B: Responder - Early Withdrawal | Treatment Phase B: Non-responder - Study Drug | Treatment Phase B: Non-responder - Standard of Care
Started | 0 (Zero participants noted because participants had completed Phase A) | 2 (Participants in this group continued treatment with the study drug) | 3 (Participants in this group did not receive additional study drug after Phase A) | 1 (Participants in this group could continue study drug treatment, per the investigator's discretion) | 1 (Participants in this group could receive the investigator's preferred standard of care)
Received At Least 1 Dose of Study Drug (Phase B Safety Sample) | 0 | 2 | 3 | 1 | 1
Completed | 0 | 2 | 3 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population - Provided following 3 core datasets used for all efficacy analyses: Treatment Phase A; Treatment Phase B responders; Treatment Phase B non-responders.
Groups:
- Treatment Phase A: During Treatment Phase A, participants received tolvaptan once daily on Days 1 and 2. If the serum sodium level did not increase at least 4 mEq/L by Day 2, treatment was extended one additional day (Day 2a). On Day 2a, participants achieving an increase in serum sodium of ≥4 mEq/L were defined as responders, and participants not achieving a ≥4 mEq/L increase in serum sodium were defined as non-responders. Participants who were responders (serum sodium increased by ≥4 mEq/L) continued to Treatment Phase B (Randomization Phase) on Day 3.
Arm/Group | Treatment Phase A
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.1 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6
  Black or African American | 1
  American Indian or Alaskan Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Change In Serum Sodium Concentration For Responders
Description: Change in serum sodium concentration (mEq/L) for responders from Day 2 (or Day 2a) at the end of Treatment Phase A (where all participants received tolvaptan) to the end of Treatment Phase B for the Early compared to Late Withdrawal groups is reported. Once a participant was randomized to Treatment Phase B, any additional therapies for the purpose of raising serum sodium, including fluid restriction, were considered rescue therapy. Upon receipt of rescue therapy, a participant's endpoint data was collected and then censored from the efficacy analysis thereafter, unless specified.
Time Frame: Day 2/2a, Day 4
Population: Treatment Phase B Responders: full analysis dataset comprised of all participants in the Phase B Safety Sample with both baseline and at least 1 postrandomization serum sodium evaluation in Phase B.
Measure: Mean (Standard Deviation); unit: mEq/L
Groups:
- Responder - Late Withdrawal: Participants who were responders (serum sodium increased by ≥4 mEq/L) from Phase A continued to Treatment Phase B (Randomization Phase) on Day 3 and were randomized to the Late Withdrawal group (continuing tolvaptan treatment for Days 3 and 4).
- Responder - Early Withdrawal: Participants who were responders (serum sodium increased by ≥4 mEq/L) from Phase A continued to Treatment Phase B (Randomization Phase) on Day 3 and were randomized to the Early Withdrawal group (not receiving additional tolvaptan on Days 3 or 4). Participants randomized to Early Withdrawal were monitored for any interventions needed to maintain appropriate serum sodium levels. Where sodium levels declined by ≥4 mEq/L, or where the overall clinical condition warranted further intervention to increase serum sodium levels, participants were treated per the investigator's preferred standard of care. Any intervention, including fluid restriction, during the first 48 hours of the Early Withdrawal phase was defined as rescue therapy, and participant data was censored thereafter.
Arm/Group | Responder - Late Withdrawal | Responder - Early Withdrawal
Number analyzed (Participants) | 2 | 3
mEq/L | -4.0 (4.2) | -1.0 (1.0)

2. Secondary Outcome: Change In Serum Sodium Concentration During Treatment Phase A
Description: Change in serum sodium concentration (mEq/L) from baseline to the end of Day 2 (or 2a) during Treatment Phase A for all participants (responders and non-responders) is reported.
Time Frame: Baseline, Day 2/2a
Population: Treatment Phase A: all participants in the Phase A Safety Sample and who had baseline and at least 1 postbaseline serum sodium evaluation in Phase A.
Measure: Mean (Standard Deviation); unit: mEq/L
Groups:
- Phase A: All Participants: During Treatment Phase A, participants received tolvaptan once daily on Days 1 and 2. If the serum sodium level did not increase at least 4 mEq/L by Day 2, treatment was extended one additional day (Day 2a). On Day 2a, participants achieving an increase in serum sodium of ≥4 mEq/L were defined as responders, and participants not achieving a ≥4 mEq/L increase in serum sodium were defined as non-responders.
Arm/Group | Phase A: All Participants
Number analyzed (Participants) | 9
mEq/L
  Day 1: 24 hours Post Dose: number analyzed (Participants) | 8
  Day 1: 24 hours Post Dose | 1 (3)
  Day 2: 24 hours Post Dose: number analyzed (Participants) | 7
  Day 2: 24 hours Post Dose | 3.4 (4.8)
  Day 2a: 24 hours Post Dose: number analyzed (Participants) | 3
  Day 2a: 24 hours Post Dose | 2.3 (2.1)

3. Secondary Outcome: Fluid Balance (Intake Minus Output) During Treatment Phase A
Description: Every 6 hours and for the 24-hour daily interval on Days 1 and 2 during Treatment Phase A, fluid balance (milliliters [mL]) was determined by fluid intake (oral and intravenous) minus urine output. Improved fluid balance would be indicated through the induction of increased urine volume. Fluid balance was monitored per institutional guidelines.
Time Frame: Every 6 hours on Days 1 and 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Phase A: All Participants
Number analyzed (Participants) | 9
mL
  Day 1: 0-6 hours | -1 (505)
  Day 1: 6-12 hours | -261 (533)
  Day 1: 12-18 hours | -36 (253)
  Day 1: 18-24 hours | 31 (344)
  Day 1: 0-24 hours | -268 (849)
  Day 2: 0-6 hours: number analyzed (Participants) | 8
  Day 2: 0-6 hours | -101 (376)
  Day 2: 6-12 hours: number analyzed (Participants) | 8
  Day 2: 6-12 hours | 6 (513)
  Day 2: 12-18 hours: number analyzed (Participants) | 8
  Day 2: 12-18 hours | -45 (400)
  Day 2: 18-24 hours: number analyzed (Participants) | 8
  Day 2: 18-24 hours | -21 (191)
  Day 2: 0-24 hours: number analyzed (Participants) | 8
  Day 2: 0-24 hours | -160 (733)

ADVERSE EVENTS:
Time Frame: From screening through early termination or follow-up phase (14 days postrandomization).
Groups:
- Treatment Phase A: During Treatment Phase A, participants received tolvaptan once daily on Days 1 and 2. If the serum sodium level did not increase at least 4 mEq/L by Day 2, treatment was extended one additional day (to Day 2a). On Day 2a, participants achieving an increase in serum sodium of ≥4 mEq/L were defined as responders, and participants not achieving a ≥4 mEq/L increase in serum sodium were defined as non-responders.
Arm/Group | Treatment Phase A | Treatment Phase B: Responder - Late Withdrawal | Treatment Phase B: Responder - Early Withdrawal | Treatment Phase B: Non-responder - Study Drug | Treatment Phase B: Non-responder - Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/2 | 0/3 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/9 | 1/2 | 0/3 | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 3/9 | 1/2 | 2/3 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase A (N=9) | Treatment Phase B: Responder - Late Withdrawal (N=2) | Treatment Phase B: Responder - Early Withdrawal (N=3) | Treatment Phase B: Non-responder - Study Drug (N=1) | Treatment Phase B: Non-responder - Standard of Care (N=1)
Catheter site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0
Medical device site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Faecal volume increased (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase A (N=9) | Treatment Phase B: Responder - Late Withdrawal (N=2) | Treatment Phase B: Responder - Early Withdrawal (N=3) | Treatment Phase B: Non-responder - Study Drug (N=1) | Treatment Phase B: Non-responder - Standard of Care (N=1)
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Issues with recruitment and enrollment made trial execution highly impracticable. This ultimately led to termination of the trial. The study was not terminated due to safety reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review, edit, and authorize publications.

DOCUMENTS (2):
  • Study Protocol (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT02012959/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT02012959/SAP_001.pdf